CLINICAL TRIAL: NCT06926114
Title: Is Microlearning the Alternative in the Age of Hyperconnectivity: A Quasi-Experimental Study
Brief Title: Is Microlearning the Alternative in the Age of Hyperconnectivity
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Medicine, Sousse (Other)
Responsible Party: Principal Investigator, Saoussen Layouni, Associate Professor, Faculty of Medicine, Sousse
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Faculty of medicine of sousse
Record Dates: First submitted 2025-03-25; First posted 2025-04-13 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-04

CONDITIONS: Knowledge Acquisition; Engagements and Motivation
Keywords: Microlearning; Medical Education; Digital Natives; Hyperconnectivity; Spinal deformities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Microlearning group (Experimental): thirteen students will be included into the microlearning group
  Interventions: Device: Microlearning intervention
- Traditional block-format module group (Active Comparator): eleven students will be included into traditional block-format module group
  Interventions: Device: Traditional block-format module group

INTERVENTIONS:
Device: Microlearning intervention — thirteen students will be included into the microlearning group will receive sequential daily learning units over ten days, . Pretest, immediate post-test, and one-month post-intervention assessments will be performed using standardized MCQ and SAQ instruments. Learner engagement, time investment, and content clarity will be additionally evaluated via structured surveys.
  Arms: Microlearning group
Device: Traditional block-format module group — eleven students will be inclued into the self block module group will engage in a comprehensive two-day self-learning module. Pretest, immediate post-test, and one-month post-intervention assessments will be performed using standardized MCQ and SAQ instruments. Learner engagement, time investment, and content clarity will be additionally evaluated via structured surveys.
  Arms: Traditional block-format module group

SUMMARY:
This Quasi-Experimental Study evaluated whether microlearning a strategy delivering brief, focused learning units enhances knowledge acquisition and retention among fifth-year medical students studying pediatric spinal deformities compared to a traditional block-format module.

Methods: twenty-four students will be included into two groups. The microlearning group will receive sequential daily learning units over ten days, while the traditional group will engage in a comprehensive two-day self-learning module. Pretest, immediate post-test, and one-month post-intervention assessments will be performed using standardized MCQ and SAQ instruments. Learner engagement, time investment, and content clarity were additionally evaluated via structured surveys.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled fifth-year medical students Registered for the optional module in Physical Medicine and Rehabilitation Access to a personal computer, tablet, or smartphone with internet connectivity Ability to access the institutional Modular Object-Oriented Dynamic Learning Environment (Moodle) learning management system (LMS) Voluntary oral informed consent Commitment to complete both pre-assessment and post-assessment evaluations Willingness to participate in either learning modality (microlearning or traditional block-format) as determined by randomization

Exclusion Criteria:

Failure to complete the pretest assessment Non-completion of the pre and post-test assessment Withdrawal of consent at any point during the study Development of circumstances that would render continued participation burdensome to the participant

Min Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-07 (Estimated)

PRIMARY OUTCOMES:
knowledge acquisition : Short and long-term retention | Immediatly post intervention score and one month post intervention score and the difference between pre and immediate post intervention score

CONTACTS AND LOCATIONS:
Locations (1):
- TUN, Sousse, Tunisia

IPD SHARING:
Plan to Share IPD: No